CLINICAL TRIAL: NCT06902636
Title: Patient Experience of Older Adults Living Alone With Injuries and Long-Term Effects of Geriatric Trauma Care Program for Living Alone Older Adults With Injuries
Brief Title: Geriatric Trauma Care Program for Living Alone Older Adults With Injuries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Santo Imanuel Tonapa, Principal investigator, Kaohsiung Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMUHIRB-F(I)-20230043; NSTC113-2314-B-037-050-MY2-1 (Other Grant/Funding Number: National Science and Technology Council of Taiwan)
Record Dates: First submitted 2025-03-21; First posted 2025-03-30 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Limb Injury; Older Adults; Geriatric; Pain; Geriatric Depression; Barthel Index; Quality of Life; Loneliness
Keywords: Limb injury; geriatric trauma; older adults; loneliness
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, two-arm experimental design will be used.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): The control group will have the routine care only
- Geriatric Trauma Care Program (Experimental): The experiment group will implement the Geriatric Trauma Care Program (GTCP) and routine care. The GTCP will be implemented through an E-book that includes six units of intervention for older adults with traumatic injuries who live alone.
  Interventions: Behavioral: Geriatric trauma care program

INTERVENTIONS:
Behavioral: Geriatric trauma care program — The experiment group will implement the Geriatric trauma care program (GTCP) and routine care. The GTCP will be implemented by a nurse practitioner and equipped with digitalized educational material, including six units of intervention for older adults with traumatic injuries who live alone.
  Arms: Geriatric Trauma Care Program

SUMMARY:
To examine the long-term effects of the Geriatric Trauma Care Program (GTCP) regarding pain, functional disability, depression, loneliness, and health-related quality of life among older adults with traumatic injuries who live alone.

DETAILED DESCRIPTION:
Traumatic injuries among older adults represent a significant public health concern due to their potential to severely affect individuals' long-term physical, emotional, and social well-being. Older adults who experience traumatic injuries often face substantial challenges during recovery, particularly those living alone who may lack sufficient support systems, exacerbating their vulnerability to chronic health issues. Pain, functional disability, depression, loneliness, and diminished health-related quality of life are prevalent adverse outcomes following traumatic injuries, underscoring the critical need for effective, targeted care strategies to address these multidimensional impacts.

The Geriatric Trauma Care Program (GTCP) is a nurse practitioner-led, digitalized trauma care program designed to provide comprehensive and accessible intervention aimed at improving immediate trauma care outcomes and facilitating sustainable recovery among older adults. While short-term benefits of digitally supported, geriatric-focused trauma interventions have been documented, the long-term effectiveness of such programs, especially for older individuals who live alone, remains less understood. Consequently, examining the enduring impact of the GTCP is essential to determine its effectiveness in fostering sustained recovery and improving quality of life for this vulnerable population. This study aims to address this gap by evaluating the long-term effects of the GTCP on pain, functional disability, depression, loneliness, and health-related quality of life among older adults with traumatic injuries who live alone. Findings from this research will provide valuable insights for healthcare providers and policymakers to enhance care delivery models, optimize resource allocation, and ultimately improve long-term outcomes for older adults recovering from traumatic injuries.

ELIGIBILITY:
Inclusion Criteria:

1. willing to join this study for three months
2. with limb injuries
3. living alone in a household
4. aged 65 years old or older
5. independent before a traumatic injury
6. having a smartphone.

Exclusion Criteria:

1. with an ISS greater than 16 (severe injuries)
2. having cognitive impairments
3. diagnosed with psychiatric illness

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Day 1 at Hospital discharge, 1 month, and 3 months
  Measured by the Numeric Pain Rating Scale with the numbers 0-10, with 0 meaning no pain and 10 meaning the worst pain.
Functional disability | Day 1 at Hospital discharge, 1 month, and 3 months
  The Barthel's Index consists of 30 items, ranging from 0 to 100, with higher scores indicating greater functional capacity.
Depression | Day 1 at Hospital discharge, 1 month, and 3 months
  The Geriatric Depression Scale Short Form, which comprises 15 items scored on a two-point scale (0 = no, 1 = yes). It scores ranged from 0-15 with the higher indicated the more severe depression symptoms.
Loneliness | Day 1 at Hospital discharge, 1 month, and 3 months
  The Elderly Loneliness Scale has eight items, with a higher score indicating more loneliness.
Health-related quality of life | Day 1 at Hospital discharge, 1 month, and 3 months
  The EuroQol-5D has five items with higher score indicated a worse health condition.

CONTACTS AND LOCATIONS:
Overall Officials: Bih-O Lee, PhD, Principal Investigator — College of Nursing, Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City, Kaohsiung, Taiwan

IPD SHARING:
Plan to Share IPD: No